CLINICAL TRIAL: NCT00844948
Title: Development of a Convenient, Automated, Objective Measure of Depression
Brief Title: Vocal Acoustic Biomarkers in Depression
Acronym: Speech2
Status: Completed | Type: Observational
Sponsor: Center for Psychological Research, Madison, WI (Other)
Collaborators: Massachusetts General Hospital (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2008P000110; 5R44MH068950-03 (NIH)
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-04

CONDITIONS: Depression
Keywords: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Young adults (18-25 years old): Young adults (18-25 years old). Major Depressive - eligible subjects will meet a baseline depression severity score of 10 or greater on the QIDS-C & QIDS-IVR, will have recently started treatment or about to start receiving treatment for MDD. Exclusion: subjects with suicidal ideation; subjects who have a history or current diagnosis of the following DSM-IV psychiatric illness: organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders not otherwise specified, bipolar disorder, patients with mood congruent or mood incongruent psychotic features, patients with substance dependence disorders, other than alcohol, active within the last 12 months; subjects with a history or current diagnosis of dementia or diagnosis or history of hypothyroidism.
- Elderly (60-80 years old): Elderly (60-80 years old). Major Depressive - eligible subjects will meet a baseline depression severity score of 10 or greater on the QIDS-C & QIDS-IVR, will have recently started treatment or about to start receiving treatment for MDD. Exclusion: subjects with suicidal ideation; subjects who have a history or current diagnosis of the following DSM-IV psychiatric illness: organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders not otherwise specified, bipolar disorder, patients with mood congruent or mood incongruent psychotic features, patients with substance dependence disorders, other than alcohol, active within the last 12 months; subjects with a history or current diagnosis of dementia or diagnosis or history of hypothyroidism.
- Chinese speakers: Chinese speakers (Mandarin or Cantonese). Major Depressive - eligible subjects will meet a baseline depression severity score of 10 or greater on the QIDS-C & QIDS-IVR, will have recently started or about to start receiving treatment for MDD. Exclusion: subjects with suicidal ideation; subjects who have a history or current diagnosis of the following DSM-IV psychiatric illness: organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders not otherwise specified, bipolar disorder, patients with mood congruent or mood incongruent psychotic features, patients with substance dependence disorders, other than alcohol, active within the last 12 months; subjects with a history or current diagnosis of dementia or diagnosis or history of hypothyroidism.

SUMMARY:
This Phase II SBIR study will replicate pilot study methods establishing computer-automated methods for assessing depression severity using interactive voice response system technology and demonstrating feasibility of obtaining measures of depression severity and treatment response through vocal acoustic analysis of speech samples obtained over the telephone. The study will automate vocal acoustic analysis methods, evaluate applicability to other patient populations (non-English speakers, children/young adult, and geriatric), and further develop multivariate acoustic models to enhance biomarker sensitivity to treatment response and prediction of the response likelihood for individual patients.

DETAILED DESCRIPTION:
This study will incorporate IVR data collection procedures developed in a prior pilot study into a multi-site industry-sponsored Phase 4 randomized, double-blind, placebo-controlled study (NCT00406952) using an established antidepressant at a therapeutically efficacious dose. The analytic procedures used to extract the vocal acoustic measures will be automated to facilitate near rapid turn around between speech sample acquisition and delivery of biomarker outcomes data. Multivariate models of vocal acoustic information to enhance the sensitivity of treatment response measurement and prediction of patient response likelihood will be further refined.

A total of 150 subjects will be recruited in the proposed studies, a sample of 50 from each of three targeted depressed patient populations - young adults (18-25 years old), elderly patients (60 years and older), and recent Asian immigrants with financial, linguistic, and cultural barriers to health care access. Eligible subjects will meet diagnostic criteria for Major Depressive Disorder, provide written informed consent, and will have baseline depression severity scores of 10 or greater on the QIDS. Pregnant women, women of child bearing potential not using a medically accepted means of contraception, suicidal or homicidal patients, or those with unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, hematological disease, or with clinical or laboratory evidence of hypothyroidism will be excluded. Patients beginning a new treatment for depression will be clinically evaluated (QIDS-C) during face-to-face interviews at the beginning of treatment (Baseline), and followed up 4 (study midpoint) and 8 weeks later (end-point). After completing the clinical interviews study participants will complete a series of IVR-based assessments using a standard desktop touch-tone telephone.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 80.
2. Written informed consent.
3. Current MDD according to the fourth version of the Diagnostic and Statistical Manual for Mental Disorders (DSM-IV)
4. Recently started to receive or about to start receiving treatment for MDD
5. Quick Inventory of Depressive Symptomatology - Clinician-Rated (QIDS-C) and QIDS-IVR scores equal or greater than 10 at baseline visit.

Exclusion Criteria:

1. Subjects with suicidal ideation where outpatient treatment is determined unsafe by the study clinician. These patients will be immediately referred to appropriate clinical treatment.
2. History or current diagnosis of the following DSM-IV psychiatric illness: organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders not otherwise specified, bipolar disorder, patients with mood congruent or mood incongruent psychotic features, patients with substance dependence disorders, other than alcohol, active within the last 12 months.
3. History or current diagnosis of dementia.
4. Diagnosis or history of hypothyroidism.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: English speaking: Young Adults, age 18-25; Elderly, age 60-80. Chinese speaking (Mandarin or Cantonese): age 18-80.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Motoric and frequency-based change in the vocal acoustic properties of speech associated with clinical improvement measured by the Quick Inventory of Depressive Symptomatology - IVR (QIDS-IVR). | baseline, week 4 & week 8

SECONDARY OUTCOMES:
Multivariate logistic regression models of vocal acoustic properties optimized for sensitivity to treatment response and prediction of the response likelihood fitted to data obtained in NCT00407952. | baseline, week 4, week 8

CONTACTS AND LOCATIONS:
Overall Officials: James C Mundt, PhD, Principal Investigator — Center for Psychological Research, Training and Consultation
Locations (2):
- United States (2):
  - South Cove Community Health, Boston, Massachusetts
  - Massachusetts General Hospital Depression Clinical and Research Program, Boston, Massachusetts